CLINICAL TRIAL: NCT04803604
Title: Decision Support Training for Advanced Cancer Family Caregivers: The CASCADE Factorial Trial
Acronym: CASCADE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James N Dionne-Odom, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01CA262039 (NIH)
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Family Members; Cancer
Keywords: family caregiver; decision-making; multiphase optimization strategy; factorial trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 2x2x2x2 full factorial pilot randomized trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collectors and principal investigator will be blind to participant condition; participants will be instructed NOT to discuss their assignment with data collectors. Trials participants will know their intervention condition as will the lay coach involved in delivering the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Basic social support + communication + Ottawa guide + 1 monthly follow up call (Experimental): 3 in-person/telephone weekly sessions on providing social support, tips for good communication, decision support tools, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + communication + Ottawa guide + monthly follow up calls for 24 weeks (Experimental): 3 in-person/telephone weekly sessions on providing social support, tips for good communication, decision support tools, and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + communication + 1 monthly follow up call (Experimental): 2 in-person/telephone weekly sessions on providing social support, tips for good communication, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + communication + monthly follow up calls for 24 weeks (Experimental): 2 in-person/telephone weekly sessions on providing social support, tips for good communication, and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + Ottawa guide + 1 monthly follow up call (Experimental): 2 in-person/telephone weekly sessions on 1 coaching session on providing social support, decision support tools, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + Ottawa guide + monthly follow up calls for 24 weeks (Experimental): 2 in-person/telephone weekly sessions on providing social support, decision support tools, and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + 1 monthly follow up call (Experimental): 1 in-person/telephone weekly sessions on providing social support and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + monthly follow up calls for 24 weeks (Experimental): 1 in-person/telephone weekly sessions on providing social support and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + communication + Ottawa guide + 1 monthly follow up call (Experimental): 5 in-person/telephone weekly sessions on providing social support, tips for good communication, decision support tools, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + communication + Ottawa guide + monthly follow up calls for 24 weeks (Experimental): 5 in-person/telephone weekly sessions on providing social support, tips for good communication, decision support tools, and monthly follow-up calls for 6
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + communication + 1 monthly follow up call (Experimental): 4 in-person/telephone weekly sessions on providing social support, tips for good communication, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + communication + monthly follow up calls for 24 weeks (Experimental): 4 in-person/telephone weekly sessions on providing social support, tips for good communication, and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + Ottawa guide + 1 monthly follow up call (Experimental): 4 in-person/telephone weekly sessions on providing social support, decision support tools, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + Ottawa guide + monthly follow up calls for 24 weeks (Experimental): 4 in-person/telephone weekly sessions on providing social support, decision support tools, and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + 1 monthly follow up call (Experimental): 3 in-person/telephone weekly sessions on providing social support, and a single monthly follow-up call
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + monthly follow up calls for 24 weeks (Experimental): 3 in-person/telephone weekly sessions on providing social support, and monthly follow-up calls for 6 months
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)

INTERVENTIONS:
Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners) — CASCADE (CAre Supporters Coached to be Adept DEcision partners) is a multicomponent, lay coach-led supportive care intervention designed to increase family caregivers' skills in providing decision support to individuals with advanced cancer. In a series of weekly, one-on-one, 15-20 minute, in-person or telephone sessions, family caregivers receive psychoeducation on principles of providing effective social support and decision partnering, decision support communication, and Ottawa Decision Guide training as well as monthly follow-up.

SUMMARY:
Using a highly innovative methodology, the Multiphase Optimization Strategy (MOST), the purpose of this randomized factorial trial is to identify components of a intervention (CASCADE) to enhance the decision support skills of family caregivers of persons with newly-diagnosed advanced cancer. Using a 2x2x2x2 full factorial design, 256 family caregivers of persons with newly-diagnosed advanced cancer will be randomized to receive one or more nurse coach-delivered decision partnering training components, based on the Ottawa Decision Support Framework and Social Support Effectiveness Theory: 1) psychoeducation on effective decision partnering principles (1 vs. 3 sessions); 2) decision partnering communication training (yes vs. no); 3) Ottawa Decision Guide training (yes vs. no); and monthly follow (1 monthly follow-up call vs. monthly follow-up calls for 24 weeks).

DETAILED DESCRIPTION:
A priority focus in oncology and palliative care is preparing the 3.2 million U.S. family caregivers of persons with cancer to effectively partner with patients in health-related decision-making from diagnosis to the end of life, particularly in underserved settings. Over 70% of patients with cancer involve relatives, friends, and partners in healthcare decisions, including choices about cancer treatments, surgery, transitions and location of care, accessing palliative and hospice care, and many others. Patients making healthcare decisions with unprepared family caregivers may experience inadequate family decision support leading to heightened distress and receipt of care/treatments inconsistent with their values and preferences. This in turn may increase distress for family caregivers. Hence, there is a critical need to train cancer family caregivers to effectively support patient decision-making; however, few interventions exist that enhance caregiver skills in providing decision support.

We have developed and successfully pilot tested CASCADE (CAre Supporters Coached to be Adept DEcision partners), a lay navigator-led, telehealth early palliative care intervention to train advanced cancer caregivers how to effectively partner with patients in health-related decision-making. Evolving out of our prior early palliative care caregiving interventions, decision partnering relevant content for family caregivers includes principles of effective social support in decision-making, decision support communication, and Ottawa Decision Guide training; however we do not know which of these components and component interactions influences patient and caregiver decision-making outcomes. Traditional research approaches typically treat interventions as "bundled" treatment packages, making it difficult to assess definitively which aspects of an intervention can be reduced, eliminated, or replaced to improve efficiency. Using traditional research methods (e.g., two-arm randomized controlled trials that test new features one at a time) requires conducting multiple studies, which is an exorbitantly expensive and time consuming process. This paradox prompts us to consider methodologies that offer a more efficient way to test multiple intervention components simultaneously. The research question we raise is: "What set of decision support training components best optimizes family caregiver support of patient healthcare decision-making?"

Using a highly innovative methodology, the Multiphase Optimization Strategy (MOST), the purpose of this study is to conduct an optimization trial to develop and refine the decision support skills of family caregivers of persons with newly-diagnosed advanced cancer (CASCADE: CAre Supporters Coached to be Adept DEcision partners). Using a 2x2x2x2 factorial design, 256 family caregivers of persons with newly-diagnosed advanced cancer will be randomized to receive one or more lay coach-delivered decision support training components, based on the Ottawa Decision Support Framework and Social Support Effectiveness Theory: 1) psychoeducation on effective decision support and social support principles (1 vs. 3 sessions); 2) decision support communication training (yes vs. no); 3) Ottawa Decision Guide training (yes vs. no); and 4) monthly follow-up (1 monthly follow-up call vs. monthly follow-up calls for 24 weeks).

The specific aims of this study are to:

Aim 1: Identify CASCADE decision support training components (main effects/interactions) that contribute meaningfully to improvement over 24 weeks in the primary outcome, patient-reported decisional conflict, measured by the Decisional Conflict Scale and secondary outcomes, including:

Caregivers: a) distress (Hospital Anxiety and Depression Scale),42 b) quality of life (PROMIS Global 10) Patients: a) distress (Hospital Anxiety and Depression Scale), b) quality of life (PROMIS Global 10), c) healthcare utilization, d) advance directive completion. A component will be considered effective if its presence produces a statistically significant main effect or two-way interaction of Cohen's d ≥.30.

Aim 2: Apply results obtained in Aim 1 to build: (1) an intervention made up of only active components and (2) a second intervention that is optimized for scalability and cost. Intervention (1) will be made up of the best set of component and component levels, based on Aim 1 results. Intervention (2) will be comprised of the set of components for the smallest cost that still yields a clinically meaningful effect in outcomes (d≥.30).

Exploratory Aim: Explore mediators and moderators (e.g., sociodemographics, decision self-efficacy, social support) of the relationship between intervention components and patient and caregiver outcomes.

ELIGIBILITY:
FAMILY CAREGIVERS

Inclusion Criteria:

1. ≥21 years of age;
2. self-endorsing or identified by the patient as "a relative, friend, or partner that has a close relationship with you and who assists you with your medical decisions and who may or may not live in the same residence as you and who is not paid for their help";
3. caring for a patient with advanced-stage cancer (see definition under Patient Inclusion criteria below);
4. caregivers will need to have an agreeable patient willing to participate in the study for data collection; and
5. English-speaking and able to complete baseline measures.

Exclusion Criteria:

1) Self-reported mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse.

PATIENTS

Inclusion Criteria:

1. ≥21 years of age;
2. diagnosed within 60 days of initial screening with an advanced cancer, defined as metastatic and/or recurrent/progressive stage III/IV cancer, including brain, lung, breast, gynecologic, head and neck, gastrointestinal, genitourinary cancer, melanoma, and hematologic malignancies.

Exclusion Criteria:

1) Medical record documentation of active severe mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient reported decisional conflict using the Decisional Conflict Scale | Baseline to 24 weeks
  16-item measure; perceptions of uncertainty in choosing options, factors contributing to uncertainty (e.g., feeling uninformed, unclear values) and feeling that decisions were informed and values-based.

SECONDARY OUTCOMES:
Patient distress as measured by the Hospital Anxiety and Depression Scale | Baseline to 24 weeks
  14 items total, 7 items measure anxiety (e.g., feeling tense, restless, worry), 7 items measure depressive symptoms (e.g., cheerfulness, feeling slowed down). Higher scores=worse anxiety/depression.
Patient quality of life as measured by the PROMIS Global Health 10 | Baseline to 24 weeks
  10 items, measures global health-related quality of life (HRQOL) in 2 domains: physical and mental health; scoring allows for estimates of cost effectiveness. Higher scores=higher HRQOL.
Patient healthcare utilization including advance directive completion as reported by family caregivers | Baseline to 24 weeks
  Inpatient days, ICU days, ED visits, urgent care visits, hospice use, palliative care provider visits, advance care planning conversations, advance directive completion, DNR orders
Caregiver distress as measured by the Hospital Anxiety and Depression Scale | Baseline to 24 weeks
  14 items total, 7 items measure anxiety (e.g., feeling tense, restless, worry), 7 items measure depressive symptoms (e.g., cheerfulness, feeling slowed down). Higher scores=worse anxiety/depression.
Caregiver quality of life as measured by the PROMIS Global Health 10 | Baseline to 24 weeks
  0 items, measures global health-related quality of life (HRQOL) in 2 domains: physical and mental health; scoring allows for estimates of cost effectiveness. Higher scores=higher HRQOL.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gazaway S, Wells RD, Azuero A, Pisu M, Guastaferro K, Rini C, Taylor R, Reed RD, Harrell ER, Bechthold AC, Bratches RW, McKie P, Lowers J, Williams GR, Rosenberg AR, Bakitas MA, Kavalieratos D, Dionne-Odom JN. Decision support training for advanced cancer family caregivers: Study protocol for the CASCADE factorial trial. Contemp Clin Trials. 2023 Aug;131:107259. doi: 10.1016/j.cct.2023.107259. Epub 2023 Jun 5. PMID 37286131